CLINICAL TRIAL: NCT07057050
Title: Constraint-induced Movement Therapy Versus Task-oriented Training
Brief Title: Constraint-induced Movement Therapy Versus Task-oriented Training On Upper Extremity Function Post-Botox Injection in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reem Hesham Mohamed Abdelhady, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Reem-Phd
Record Dates: First submitted 2025-06-28; First posted 2025-07-09 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Constraint Induced Movement Therapy; Task Oriented Training; Botox Injection; Upper Extremity Function; Stroke
MeSH Terms: conditions — Stroke | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- constrained induced movement therapy (Experimental): Patients will undergo a 60-minute physiotherapy program, such as traditional upper extremity training, following botulinum toxin A injection, as well as constrained induced movement therapy tasks for 12 consecutive weeks.
  Interventions: Other: The designed physiotherapy program; Drug: The Botulinum toxin injection; Other: Constrained induced movement therapy
- task-oriented training (Active Comparator): Patients will undergo a 60-minute physiotherapy program, such as traditional upper extremity training, following botulinum toxin A injection, as well as task-oriented training tasks for 12 consecutive weeks.
  Interventions: Other: The designed physiotherapy program; Drug: The Botulinum toxin injection; Other: Task oriented training
- designed physical therapy program (Active Comparator): Patients will undergo a 60-minute physiotherapy program, such as traditional upper extremity training, following botulinum toxin A injection, for 12 consecutive weeks.
  Interventions: Other: The designed physiotherapy program; Drug: The Botulinum toxin injection

INTERVENTIONS:
Other: The designed physiotherapy program — * Scapular and thoracic mobilization, active assisted and passive exercises, and positioning such as weight bearing on the affected upper limb.
  * Strengthening of the shoulder flexors and elbow and wrist extensors.
  * Stretching exercises of the spastic muscles (shoulder extensors, elbow and wrist flexors.)
Drug: The Botulinum toxin injection — The injection of 1000 units per upper extremity will be done into the biceps brachii muscle at 2 sites, and 150 units into the flexor carpi radialis muscle at 1 site per muscle, using anatomical landmarks similar to routine electromyography.
Other: Task oriented training — The training involves 30 minutes of bilateral functional tasks like carrying a block, grabbing and folding a towel, staking cups upright, holding a glass and drinking water, throwing a ball into a basket, and moving pegs.
  Arms: task-oriented training
Other: Constrained induced movement therapy — The therapy session focuses on enhancing the affected arm's functional tasks, such as throwing a ball, holding a glass, combing hair, turning on and off a light switch, grasping and releasing blocks, pouring from glass to another, moving cups, and moving pegs. Participants are instructed to wear a restrictive mitt on their non-paretic hand for 6 hours a day for 4 days, 7 weeks, and 12 weeks, with the mitt removed for safety, hygiene, or agreed-on activities.
  Arms: constrained induced movement therapy

SUMMARY:
This study will be conducted to determine the impact of Constraint-Induced Movement Therapy versus Task-Oriented Training on upper extremity function post-Botox injection in stroke patients.

DETAILED DESCRIPTION:
Arm and hand movement problems are significant contributors to disability in stroke patients, with only 5% regaining full arm function and 20% regaining no functional use. Alternative strategies are needed to reduce long-term disability and upper limb impairment in hemiparesis patients. Previous studies have used various treatment methods, including botulinum toxin, but the degree of motor improvement depends on task complexity. Future research should focus on adjunct therapy, such as task-specific training and constrained induced therapy, in addition to botulinum toxin treatments, to facilitate functional improvement in spastic upper extremity.

ELIGIBILITY:
Inclusion Criteria:

* The study focuses on patients aged 45-60 years
* Patients who have subacute spastic hemiplegia with occlusion of the middle cerebral artery
* Patients who are able to maintain balance in sitting positions.
* Patients are diagnosed with the affected upper extremity being the dominant side.
* Physiotherapy sessions are initiated 3-7 days post-injection,
* Patients have pre-injection Modified Ashworth scores equal to 2 (moderate spasticity) in wrist or elbow flexors.
* Patients can actively extend joints at least 10° at metacarpophalangeal and interphalangeal joints and 20° at the wrist of the affected upper limb.

Exclusion Criteria:

* Joint immobility in the upper limb due to contracture, bony deformity, or heterotopic ossification
* Significant cognitive deficits (Mini-Mental Status Examination score <24).

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
assessment of change of arm motor impairment | at baseline and after 12 weeks
  The Fugl-Meyer Upper Extremity scale, validated and reliable, correlates well with upper extremity coordination. It includes four motor sub-items relevant to the affected upper limb: shoulder/elbow/forearm, wrist, hand, and speed/coordination. The test is conducted pre- and post-treatment, requiring volitional movement mixing synergies. The total Fugl-Meyer Upper Extremity scale takes 30-35 minutes, and items are scored using a 3-point ordinal scale. The patient's performance ranges from 0 to 2 on the scale.

SECONDARY OUTCOMES:
Evaluation of degree of spasticity | at baseline and after 12 weeks
  The Modified Ashworth Scale is a 6-point scale used to measure spasticity in the affected upper limb. The score ranges from 0 to 4, with lower scores indicating normal muscle tone and higher scores indicating spasticity or increased resistance to passive movement. Muscle tone assessment is done in a comfortable, quiet room, with no nociceptive or exteroceptive stimuli. The patient is instructed to empty their bladder and release tight clothes before the assessment.
assessment of change of handgrip strength | at baseline and after 12 weeks
  Maximal voluntary grip forces (MVGF) will be assessed using grip dynamometer. Subjects are seated in a wheelchair. The shoulder is placed at approximately 30 degrees of abduction and 0 degrees of flexion. The elbow is flexed at 90 degrees with the wrist in neutral position. Maximal voluntary grip forces are established as the highest values recorded during three maximal voluntary exertions separated by 2-minute rest intervals. The mean value for each hand was used for analysis
assessment of change of shoulder and elbow movement | at baseline and after 12 weeks
  Kinovea software is a reliable method for measuring shoulder joint position sense, suitable for medical, rehabilitation, and sports environments. It accurately measures shoulder joint position up to 5 meters from an object and 90°-45° angle. Kinovea software also performs motion analysis, capturing shoulder flexion, abduction, elbow flexion, and extension movements. Cross marks are drawn on anatomical landmarks on the dominant upper limb.
assessment of change of upper limb function | at baseline and after 12 weeks
  The Action Research Arm Test (ARAT) is a tool used to evaluate limb function in individuals with hemiplegia due to cortical damage. It measures a client's ability to handle objects of different sizes, weights, and shapes. The ARAT scores range from 0 to 57, with higher scores indicating better performance. The test is conducted pre- and post-treatment and consists of four subscales: grasp, grip, pinch, and gross movement. If a client fails on the most difficult task, the easiest task is performed, and the entire subscale is scored as zero.

CONTACTS AND LOCATIONS:
Locations (1):
- outpatient clinics of Mansoura university hospital, Al Mansurah, Egypt